CLINICAL TRIAL: NCT06254729
Title: Study on the Application of Multi-omics in the Assessment of Efficacy and Prediction of Side Effects in Cervical Cancer
Brief Title: Clinical Study on the Evaluation of the Efficacy of Cervical Cancer
Acronym: EECC
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Gansu Maternal and Child Health Hospital (Unknown); Hanzhong Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YXJLRH2022039
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, urine, feces, intestinal flora
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group: The training group is used to train the model.
  Interventions: Other: Observational study
- validation group: The validation group is used to evaluate model performance.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Our study does not have any exposure factors.

SUMMARY:
The main objectives of this study are to construct a multi-omics-based prognostic and side-effect prediction model for cervical cancer based on pre-treatment imaging, digital pathology, genomics, proteomics, molecular biology, metabolomics, and intestinal flora characteristics data of cervical cancer patients, combined with patients' clinical information, to guide the precise treatment of cervical cancer patients; and to deeply excavate the characteristics related to recurrent cervical cancer based on time-series multi-omics data. Construct an artificial intelligence auxiliary model for dynamic monitoring of cervical cancer recurrence based on longitudinal multi-omics. To provide a real-time and timely tool for clinical early prediction, early identification, early diagnosis and early intervention of cervical cancer, to prolong the survival time and improve the quality of patients' survival.

1. To realize multi-omics feature extraction of cervical cancer patients before treatment, and build a prognosis and side-effect prediction model of cervical cancer to guide accurate treatment;
2. To make iterative, comprehensive, real-time assessment of the risk of recurrence of cervical cancer based on time-series multi-omics data, and to build an early warning model for early identification and early diagnosis of recurrent cervical cancer;
3. To establish a prognostic and side-effect prediction and risk dynamic assessment model for cervical cancer, to build an intelligent decision support system, to implement the application of prognostic and side-effect prediction and dynamic monitoring model, to further assist in the precise diagnosis and treatment of cervical cancer, and to provide an accurate prognostic tool for identifying, diagnosing, and intervening in cervical cancer during the follow-up process.

DETAILED DESCRIPTION:
1. Construct a prognosis and side effect prediction model based on pre-treatment multi-omics features of cervical cancer patients.

1. Case selection: According to the overall experimental design, 2800 patients in the training group were used as the training data set, and 1200 patients in the validation group were used as the validation data collection.
2. Model training and tuning: a. Extract the multi-omics features of the training group, carry out self-learning of the features, and form a preliminary cervical cancer prognosis and side-effect prediction model; b. Input the multi-omics data of the validation group into the model, and carry out the structure of the model and the training parameters, and seek for the optimal model structure and training parameters; c. Determine the optimal cervical cancer prognosis prediction and side-effect model.

2.Mining recurrent tumor characteristics based on multi-omics data and constructing a comprehensive assessment model for recurrence risk .

1. Case selection: In accordance with the overall experimental design, 2800 patients in the training group were used as the training dataset, and 1200 patients in the validation group were collected as the validation data.
2. Model training and tuning: a. The multi-omics data features of the training group before the diagnosis of recurrence in previous follow-up visits are used to carry out self-learning of the features, assess the risk of tumor recurrence based on multi-omics features in the course of previous follow-up visits, form a dynamic, real-time recurrence risk assessment model, and derive a comprehensive risk value for the decision-making of recurrence intervention; b. Multi-omics features related to the previous follow-up visits of the validation group before the diagnosis of recurrence are inputted into the model, and the iterative time-series recurrence risk assessment is carried out on the patients. time-series recurrence risk iterative assessment of patients to assess the diagnostic performance of the model; c. Adjust the structure and training parameters of the model according to the segmentation accuracy of the validation group to seek the optimal model structure and training parameters; d. Use technical means such as data augmentation and other technical means to think of enlarging the sample size to improve the segmentation accuracy; e. Determine the optimal risk assessment model.

3. Establish the prognosis and side-effect prediction and dynamic monitoring system of cervical cancer.

a. Docking the above constructed model with the outpatient system to construct a prognosis and side reaction prediction and dynamic monitoring system in the process of cervical cancer diagnosis and treatment; b. Constructing an intelligent decision support system through the prognosis and side reaction prediction and risk dynamic assessment model, implementing the application of recurrence prediction and dynamic monitoring system, and assisting the clinicians to make decisions on intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* Pathology: patients with pathologically confirmed cervical cancer
* Location: primary tumor of the cervix

Exclusion Criteria:

* Patients with no prior radiation therapy
* Patients without treatment
* Patients without regular follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients receiving radiotherapy
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-02-16 (Estimated); Primary Completion 2029-02-16 (Estimated); Study Completion 2030-02-16 (Estimated)

PRIMARY OUTCOMES:
Number of Circulating Tumor Cell Count | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Number of Circulating Tumor Cell Count (CTC count), cells/mL
Concentration of Alpha-fetoprotein (AFP) | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Concentration of Alpha-fetoprotein (AFP), ng/mL
Concentration of Carcinoembryonic Antigen (CEA) | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Concentration of Carcinoembryonic Antigen (CEA), ng/mL
Concentration of carbohydrate antigen 199 (CA199) | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Concentration of carbohydrate antigen 199 (CA199), U/mL
Concentration of Squamous Epithelial Cell Carcinoma Antigen (SCC-Ag) | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Concentration of Squamous Epithelial Cell Carcinoma Antigen (SCC-Ag), ng/mL
Concentration of carbohydrate antigen 125(CA125) | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Concentration of carbohydrate antigen 125(CA125), U/mL.
Count of Bacteria in urine | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Count of Bacteria in urine, colony-forming units (CFU)/mL.
Count of bacteria in stool | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Count of bacteria in stool, colony-forming units (CFU)/mL
5-year overall survival rate of Participants | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  the proportion of patients who are alive at least 5 years after their initial diagnosis of cancer, regardless of the cause of death,%
disease-free survival of Participants | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  the length of time from the start of treatment until either the recurrence of cancer or death from any cause, months
progression-free survival of Participants | From data of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  the start of treatment until either the recurrence of cancer or death from any cause, months

CONTACTS AND LOCATIONS:
Overall Officials: Jinlu Ma, Study Chair — First Affiliated Hospital of Xian Jiaotong University

IPD SHARING:
Plan to Share IPD: No